CLINICAL TRIAL: NCT03856996
Title: A Phase 1 Double-blind, Randomized, Controlled Clinical Trial in Healthy, HIV-1-Uninfected Adult Participants to Compare the Safety, Tolerability and Immunogenicity of CH505TF gp120 Produced From Stably Transfected Cells to CH505TF gp120 Produced From Transiently Transfected Cells
Brief Title: A Clinical Trial in Healthy, HIV-1-Uninfected Adult Participants to Compare the Safety, Tolerability and Immunogenicity of CH505TF gp120 Produced From Stably Transfected Cells to CH505TF gp120 Produced From Transiently Transfected Cells
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HVTN 123; 34569 (Registry Identifier: DAIDS-ES Registry Number)
Record Dates: First submitted 2019-02-14; First posted 2019-02-27 (Actual); Results first posted 2022-07-11 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-04

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1: Stable CH505TF gp120 + GLA-SE (Experimental): Participants in Group 1 will receive 100 mcg of Stable CH505TF gp120 admixed with 10 mcg of GLA-SE by intramuscular (IM) injection at Months 0, 2, and 6.
  Interventions: Biological: Stable CH505TF gp120; Biological: Glucopyranosyl Lipid Adjuvant-Stable Emulsion (GLA-SE)
- Group 2: Transient CH505TF gp120 + GLA-SE (Experimental): Participants in Group 2 will receive 100 mcg of Transient CH505TF gp120 admixed with 10 mcg of GLA-SE by IM injection at Months 0, 2, and 6.
  Interventions: Biological: Transient CH505TF gp120; Biological: Glucopyranosyl Lipid Adjuvant-Stable Emulsion (GLA-SE)

INTERVENTIONS:
Biological: Stable CH505TF gp120 — Administered by IM injection in the deltoid of the non-dominant arm
  Arms: Group 1: Stable CH505TF gp120 + GLA-SE
Biological: Transient CH505TF gp120 — Administered by IM injection in the deltoid of the non-dominant arm
  Arms: Group 2: Transient CH505TF gp120 + GLA-SE
Biological: Glucopyranosyl Lipid Adjuvant-Stable Emulsion (GLA-SE) — Admixed with Stable CH505TF gp120 or Transient CH505TF gp120 for IM injection in the deltoid of the non-dominant arm

SUMMARY:
The purpose of this study is to compare the safety, tolerability, and immunogenicity of CH505TF gp120 produced from stably transfected cells to CH505TF gp120 produced from transiently transfected cells in healthy, HIV-1-uninfected adult participants.

DETAILED DESCRIPTION:
This study will compare the safety, tolerability, and immunogenicity of two experimental HIV vaccines in healthy, HIV-1-uninfected adult participants. The study vaccines are called Stable CH505TF gp120 and Transient CH505TF gp120. The vaccines are mixed with an adjuvant called GLA-SE.

Participants will be randomly assigned to two groups. Participants in Group 1 will receive Stable CH505TF gp120; participants in Group 2 will receive Transient CH505TF. Depending on their group, participants will receive Stable CH505TF gp120 or Transient CH505TF gp120 by injection at Months 0, 2, and 6.

Additional study visits will occur at Months 0.5, 2.5, 6.5, 9, and 12. Study visits may include physical examinations, medical history, vaccine injections, blood and urine collection, risk reduction counseling, and questionnaires. Participants will also be contacted for health information at Month 18.

ELIGIBILITY:
Inclusion Criteria:

General and Demographic Criteria

* Age of 18 to 50 years
* Access to a participating HIV Vaccine Trials Network (HVTN) clinical research site (CRS) and willingness to be followed for the planned duration of the study
* Ability and willingness to provide informed consent
* Assessment of understanding: volunteer demonstrates understanding of this study; completes a questionnaire prior to first vaccination with verbal demonstration of understanding of all questionnaire items answered incorrectly
* Willing to be contacted in person or by phone, text message, or e-mail 6 months after completion of the scheduled clinic visits
* Agrees not to enroll in another study of an investigational research agent before the last required protocol clinic visit
* Good general health as shown by medical history, physical exam, and screening laboratory tests

HIV-Related Criteria

* Willingness to receive HIV test results
* Willingness to discuss HIV infection risks and amenable to HIV risk reduction counseling
* Assessed by the clinic staff as being at "low risk" for HIV infection and committed to maintaining behavior consistent with low risk of HIV exposure through the last required protocol clinic visit. (see study protocol)

Laboratory Inclusion Values

Hemogram/Complete blood count (CBC)

* Hemoglobin greater than or equal to 11.0 g/dL for volunteers who were assigned female sex at birth, greater than or equal to 13.0 g/dL for volunteers who were assigned male sex at birth. For transgender participants who have been on hormone therapy for more than 6 consecutive months, determine hemoglobin eligibility based on the gender with which they identify (ie, a transgender female who has been on hormone therapy for more than 6 consecutive months should be assessed for eligibility using the hemoglobin parameters for persons assigned female sex at birth).
* White blood cell count equal to 3,300 to 12,000 cells/mm^3
* Total lymphocyte count greater than or equal to 800 cells/mm^3
* Remaining differential either within institutional normal range or with site physician approval
* Platelets equal to 125,000 to 550,000/mm^3

Chemistry

* Chemistry panel: alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase less than 1.25 times the institutional upper limit of normal; creatinine less than or equal to institutional upper limit of normal.

Virology

* Negative HIV-1 and -2 blood test: US volunteers must have a negative US Food and Drug Administration (FDA)-approved enzyme immunoassay (EIA).
* Negative Hepatitis B surface antigen (HBsAg)
* Negative anti-Hepatitis C virus antibodies (anti-HCV), or negative HCV polymerase chain reaction (PCR) if the anti-HCV is positive

Urine

* Normal urine:

  * Negative urine glucose, and
  * Negative or trace urine protein, and
  * Negative or trace urine hemoglobin (if trace hemoglobin is present on dipstick, a microscopic urinalysis with red blood cells levels within institutional normal range).

Reproductive Status

* Volunteers who were assigned female sex at birth: negative serum or urine beta human chorionic gonadotropin (β-HCG) pregnancy test performed prior to vaccination on the day of initial vaccination. Persons who are NOT of reproductive potential due to having undergone total hysterectomy or bilateral oophorectomy (verified by medical records), are not required to undergo pregnancy testing.
* Reproductive status: A volunteer who was assigned female sex at birth must:

  * Agree to use effective contraception for sexual activity that could lead to pregnancy from at least 21 days prior to enrollment until 3 months after the final study vaccination. Effective contraception is defined as using the following methods:

    * Condoms (male or female) with or without a spermicide,
    * Diaphragm or cervical cap with spermicide,
    * Intrauterine device (IUD),
    * Hormonal contraception, or
    * Any other contraceptive method approved by the HVTN 123 Protocol Safety Review Team (PSRT)
    * Successful vasectomy in any partner assigned male sex at birth (considered successful if a volunteer reports that a male partner has [1] documentation of azoospermia by microscopy, or [2] a vasectomy more than 2 years ago with no resultant pregnancy despite sexual activity post vasectomy);
  * Or not be of reproductive potential, such as having reached menopause (no menses for 1 year) or having undergone hysterectomy, bilateral oophorectomy, or tubal ligation;
  * Or be sexually abstinent.
* Volunteers who were assigned female sex at birth must also agree not to seek pregnancy through alternative methods, such as artificial insemination or in vitro fertilization until after the last required protocol clinic visit

Exclusion Criteria

General

* Blood products received within 120 days before first vaccination
* Investigational research agents received within 30 days before first vaccination
* Body mass index (BMI) greater than or equal to 40; or BMI greater than or equal to 35 with 2 or more of the following: age greater than 45, systolic blood pressure greater than 140 mm Hg, diastolic blood pressure greater than 90 mm Hg, current smoker, known hyperlipidemia
* Intent to participate in another study of an investigational research agent or any other study that requires non-HVTN HIV antibody testing during the planned duration of the HVTN 123 study
* Pregnant or breastfeeding
* Active duty and reserve US military personnel

Vaccines and other Injections

* HIV vaccine(s) received in a prior HIV vaccine trial. For volunteers who have received control/placebo in an HIV vaccine trial, the HVTN 123 PSRT will determine eligibility on a case-by-case basis.
* Previous receipt of monoclonal antibodies (mAbs), whether licensed or investigational; the HVTN 123 PSRT will determine eligibility on a case-by-case basis.
* Non-HIV experimental vaccine(s) received within the last 5 years in a prior vaccine trial. Exceptions may be made by the HVTN 123 PSRT for vaccines that have subsequently undergone licensure by the FDA. For volunteers who have received control/placebo in an experimental vaccine trial, the HVTN 123 PSRT will determine eligibility on a case-by-case basis. For volunteers who have received an experimental vaccine(s) greater than 5 years ago, eligibility for enrollment will be determined by the HVTN 123 PSRT on a case-by-case basis.
* Live attenuated vaccines received within 30 days before first vaccination or scheduled within 14 days after injection (eg, measles, mumps, and rubella [MMR]; oral polio vaccine [OPV]; varicella; yellow fever)
* Any vaccines that are not live attenuated vaccines and were received within 14 days prior to first vaccination (eg, tetanus, pneumococcal, Hepatitis A or B)
* Allergy treatment with antigen injections within 30 days before first vaccination or that are scheduled within 14 days after first vaccination

Immune System

* Immunosuppressive medications received within 168 days before first vaccination (Not exclusionary: [1] corticosteroid nasal spray; [2] inhaled corticosteroids; [3] topical corticosteroids for mild, uncomplicated dermatitis; or [4] a single course of oral/parenteral prednisone or equivalent at doses less than or equal to 60 mg/day and length of therapy less than 11 days with completion at least 30 days prior to enrollment)
* Serious adverse reactions to vaccines including history of anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema, and/or abdominal pain. (Not excluded from participation: a volunteer who had a nonanaphylactic adverse reaction to pertussis vaccine as a child.)
* Immunoglobulin received within 60 days before first vaccination
* Autoimmune disease
* Immunodeficiency

Clinically significant medical conditions

* Clinically significant medical condition, physical examination findings, clinically significant abnormal laboratory results, or past medical history with clinically significant implications for current health. A clinically significant condition or process includes but is not limited to:

  * A process that would affect the immune response,
  * A process that would require medication that affects the immune response,
  * Any contraindication to repeated injections or blood draws,
  * A condition that requires active medical intervention or monitoring to avert grave danger to the volunteer's health or well-being during the study period,
  * A condition or process for which signs or symptoms could be confused with reactions to vaccine, or
  * Any condition specifically listed among the exclusion criteria below.
* Any medical, psychiatric, occupational, or other condition that, in the judgment of the investigator, would interfere with, or serve as a contraindication to, protocol adherence, assessment of safety or reactogenicity, or a volunteer's ability to give informed consent
* Psychiatric condition that precludes compliance with the protocol. Specifically excluded are persons with psychoses within the past 3 years, ongoing risk for suicide, or history of suicide attempt or gesture within the past 3 years.
* Current anti-tuberculosis (TB) prophylaxis or therapy
* Asthma exclusion criteria: Asthma other than mild, well-controlled asthma. (Symptoms of asthma severity as defined in the most recent National Asthma Education and Prevention Program (NAEPP) Expert Panel report).
* Exclude a volunteer who:

  * Uses a short-acting rescue inhaler (typically a beta 2 agonist) daily, or
  * Uses moderate/high dose inhaled corticosteroids, or
  * In the past year has either of the following:

    * Greater than 1 exacerbation of symptoms treated with oral/parenteral corticosteroids;
    * Needed emergency care, urgent care, hospitalization, or intubation for asthma.
* Diabetes mellitus type 1 or type 2 (Not excluded: type 2 cases controlled with diet alone or a history of isolated gestational diabetes.)
* Thyroidectomy, or thyroid disease requiring medication during the last 12 months
* Hypertension:

  * If a person has been found to have elevated blood pressure or hypertension during screening or previously, exclude for blood pressure that is not well controlled. Well-controlled blood pressure is defined as consistently less than or equal to 140 mm Hg systolic and less than or equal to 90 mm Hg diastolic, with or without medication, with only isolated, brief instances of higher readings, which must be less than or equal to 150 mm Hg systolic and less than or equal to 100 mm Hg diastolic. For these volunteers, blood pressure must be less than or equal to 140 mm Hg systolic and less than or equal to 90 mm Hg diastolic at enrollment.
  * If a person has NOT been found to have elevated blood pressure or hypertension during screening or previously, exclude for systolic blood pressure greater than or equal to 150 mm Hg at enrollment or diastolic blood pressure greater than or equal to 100 mm Hg at enrollment.
* Bleeding disorder diagnosed by a doctor (eg, factor deficiency, coagulopathy, or platelet disorder requiring special precautions)
* Malignancy (Not excluded from participation: Volunteer who has had malignancy excised surgically and who, in the investigator's estimation, has a reasonable assurance of sustained cure, or who is unlikely to experience recurrence of malignancy during the period of the study)
* Seizure disorder: History of seizure(s) within past three years. Also exclude if volunteer has used medications in order to prevent or treat seizure(s) at any time within the past 3 years.
* Asplenia: any condition resulting in the absence of a functional spleen
* History of hereditary angioedema, acquired angioedema, or idiopathic angioedema.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-05-23 (Actual); Primary Completion 2021-03-16 (Actual); Study Completion 2021-09-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Greg Wilson, Study Chair — Vanderbilt Medical Center; Colleen Kelley, Study Chair — Emory University
Locations (3):
- United States (3):
  - The Hope Clinic of the Emory Vaccine Center CRS, Decatur, Georgia
  - Brigham and Women's Hospital Vaccine CRS (BWH VCRS), Boston, Massachusetts
  - Vanderbilt Vaccine (VV) CRS, Nashville, Tennessee

REFERENCES:
- [Derived] Wilson GJ, Church LWP, Kelley CF, Robinson ST, Lu Y, Furch BD, Fong Y, Paez CA, Yacovone M, Jacobsen T, Maughan M, Martik D, Heptinstall JR, Zhang L, Montefiori DC, Tomaras GD, Kublin JG, Corey L. HVTN 123: A Phase 1, Randomized Trial Comparing Safety and Immunogenicity of CH505TF gp120 Produced by Stably and Transiently Transfected Cell Lines. J Infect Dis. 2025 Apr 15;231(4):e764-e769. doi: 10.1093/infdis/jiae558. PMID 39671174
- [Derived] Wolfe LS, Smedley JG 3rd, Bubna N, Hussain A, Harper R, Mostafa S. Development of a platform-based approach for the clinical production of HIV gp120 envelope glycoprotein vaccine candidates. Vaccine. 2021 Jun 29;39(29):3852-3861. doi: 10.1016/j.vaccine.2021.05.073. Epub 2021 Jun 4. PMID 34099325

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Vaccine: 100 mcg of Stable CH505TF gp120 admixed with 10 mcg of GLA-SE, to be administered as a 1mL IM injection in the deltoid of the non-dominant arm at months 0, 2, and 6
- Group 2: Vaccine: 100 mcg of Transient CH505TF gp120 admixed with 10 mcg of GLA-SE, to be administered as a 1mL IM injection in the deltoid of the non-dominant arm at months 0, 2 and 6
Period: Overall Study
Arm/Group | Group 1: Vaccine | Group 2: Vaccine
Started | 15 | 15
Completed | 12 | 13
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 1: Vaccine: 100 mcg of Stable CH505TF gp120 admixed with 10 mcg of GLA-SE, to be administered as a 1mL IM injection in the deltoid of the non-dominant arm at months 0, 2 and 6
- Total: Total of all reporting groups
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Median (Full Range); unit: years] | 28 [22 to 48] | 28 [19 to 46] | 28 [19 to 48]
Age, Customized [Count of Participants; unit: Participants]
  Less than 18 years | 0 | 0 | 0
  18 - 20 years | 0 | 2 | 2
  21 - 30 years | 11 | 8 | 19
  31 - 40 years | 3 | 3 | 6
  41 - 50 years | 1 | 2 | 3
  Above 50 years | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 7 | 7 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 15 | 13 | 28
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 14 | 13 | 27
  More than one race | 0 | 0 | 0
  Other | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Local Reactogenicity Signs and Symptoms: Pain and/or Tenderness
Description: Graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1 [July 2017]. The maximum grade observed for each symptom over the time frame is presented.
Time Frame: Measured through 7 days after each vaccine dose
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Vaccine | Group 2: Vaccine
Number analyzed (Participants) | 15 | 15
Participants
  None | 2 | 2
  Mild | 9 | 12
  Moderate | 4 | 1
  Severe | 0 | 0
  Potentially Life-threatening | 0 | 0

2. Primary Outcome: Number of Participants Reporting Local Reactogenicity Signs and Symptoms: Erythema and/or Induration
Description: as for outcome 1
Time Frame: Measured through 7 days after each vaccine dose
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Vaccine | Group 2: Vaccine
Number analyzed (Participants) | 15 | 15
Participants
  Erythema/Redness: None | 12 | 15
  Erythema/Redness: Not gradable | 0 | 0
  Erythema/Redness: Gr 1: 2.5 to less than 5 cm dim. | 0 | 0
  Erythema/Redness: Gr 2: 5 to less than 10 cm dim. | 3 | 0
  Erythema/Redness: Gr 3: >= 10cm dim. | 0 | 0
  Erythema/Redness: Gr 3: complications AE | 0 | 0
  Erythema/Redness: Gr 4: complications AE | 0 | 0
  Induration/Swelling: None | 14 | 14
  Induration/Swelling: Not gradable | 0 | 0
  Induration/Swelling: Gr 1: 2.5 to less than 5 cm dim. | 0 | 0
  Induration/Swelling: Gr 2: 5 to less than 10 cm dim. | 1 | 1
  Induration/Swelling: Gr 3: >= 10cm dim. | 0 | 0
  Induration/Swelling: Gr 3: complications AE | 0 | 0
  Induration/Swelling: Gr 4: complications AE | 0 | 0
  Erythema and/or Induration: None | 12 | 14
  Erythema and/or Induration: Not gradable | 0 | 0
  Erythema and/or Induration: Gr 1: 2.5 to less than 5 cm dim. | 0 | 0
  Erythema and/or Induration: Gr 2: 5 to less than 10 cm dim. | 3 | 1
  Erythema and/or Induration: Gr 3: >= 10cm dim. | 0 | 0
  Erythema and/or Induration: Gr 3: complications AE | 0 | 0
  Erythema and/or Induration: Gr 4: complications AE | 0 | 0

3. Primary Outcome: Number of Participants Reporting Systemic Reactogenicity Signs and Symptoms
Description: as for outcome 1
Time Frame: Measured through 7 days after each vaccine dose
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Vaccine | Group 2: Vaccine
Number analyzed (Participants) | 15 | 15
Participants
  Malaise and/or fatigue: None | 9 | 7
  Malaise and/or fatigue: Mild | 3 | 7
  Malaise and/or fatigue: Moderate | 3 | 1
  Malaise and/or fatigue: Severe | 0 | 0
  Malaise and/or fatigue: Potentially Life-threatening | 0 | 0
  Myalgia: None | 12 | 11
  Myalgia: Mild | 1 | 3
  Myalgia: Moderate | 2 | 1
  Myalgia: Severe | 0 | 0
  Myalgia: Potentially Life-threatening | 0 | 0
  Headache: None | 9 | 9
  Headache: Mild | 4 | 4
  Headache: Moderate | 2 | 2
  Headache: Severe | 0 | 0
  Headache: Potentially Life-threatening | 0 | 0
  Nausea: None | 13 | 13
  Nausea: Mild | 2 | 1
  Nausea: Moderate | 0 | 1
  Nausea: Severe | 0 | 0
  Nausea: Potentially Life-threatening | 0 | 0
  Chills: None | 13 | 14
  Chills: Mild | 2 | 0
  Chills: Moderate | 0 | 1
  Chills: Severe | 0 | 0
  Chills: Potentially Life-threatening | 0 | 0
  Arthralgia: None | 13 | 13
  Arthralgia: Mild | 1 | 2
  Arthralgia: Moderate | 1 | 0
  Arthralgia: Severe | 0 | 0
  Arthralgia: Potentially Life-threatening | 0 | 0
  Max. Systemic Symptoms: None | 6 | 5
  Max. Systemic Symptoms: Mild | 5 | 7
  Max. Systemic Symptoms: Moderate | 4 | 3
  Max. Systemic Symptoms: Severe | 0 | 0
  Max. Systemic Symptoms: Potentially Life-threatening | 0 | 0
  Temperature: None | 14 | 15
  Temperature: Mild | 0 | 0
  Temperature: Moderate | 1 | 0
  Temperature: Severe | 0 | 0
  Temperature: Potentially Life-threatening | 0 | 0

4. Primary Outcome: Chemistry and Hematology Laboratory Measures - Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Alkaline Phosphatase (ALP) in U/L
Description: For each local laboratory measure, summary statistics were presented by treatment group and timepoint for the overall population.
Time Frame: Measured during screening, Days 14, 70, 182, 273
Population: Overall Number of Participants Analyzed represents participants enrolled and eligible for laboratory assessment. Participants do not have laboratory assessments if they attended the visit but laboratory specimens were not collected, missed the scheduled visit, or terminated participation in the study prior to the scheduled visit.
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | Group 1: Vaccine | Group 2: Vaccine
Number analyzed (Participants) | 15 | 15
U/L
  Alanine Aminotransferase -Baseline | 22 [17 to 31] | 19 [14 to 25]
  Alanine Aminotransferase -Day 14 | 20 [13 to 26] | 17 [10 to 21]
  Alanine Aminotransferase -Day 70: number analyzed (Participants) | 12 | 13
  Alanine Aminotransferase -Day 70 | 18.5 [15.5 to 29] | 18 [12 to 23]
  Alanine Aminotransferase -Day 182: number analyzed (Participants) | 13 | 14
  Alanine Aminotransferase -Day 182 | 17 [14 to 20] | 18.5 [12 to 24]
  Alanine Aminotransferase -Day 273: number analyzed (Participants) | 13 | 13
  Alanine Aminotransferase -Day 273 | 17 [11 to 21] | 19 [16 to 23]
  Aspartate Aminotransferase -Baseline | 25 [19 to 27] | 19 [14 to 22]
  Aspartate Aminotransferase -Day 14 | 18 [16 to 23] | 18 [12 to 23]
  Aspartate Aminotransferase -Day 70: number analyzed (Participants) | 12 | 13
  Aspartate Aminotransferase -Day 70 | 18 [15 to 34] | 21 [16 to 24]
  Aspartate Aminotransferase -Day 182: number analyzed (Participants) | 13 | 14
  Aspartate Aminotransferase -Day 182 | 16 [13 to 24] | 21.5 [16 to 23]
  Aspartate Aminotransferase -Day 273: number analyzed (Participants) | 13 | 13
  Aspartate Aminotransferase -Day 273 | 16 [14 to 23] | 24 [17 to 28]
  Alkaline Phosphatase -Baseline | 61 [49 to 75] | 60 [50 to 67]
  Alkaline Phosphatase -Day 14 | 58 [54 to 76] | 60 [51 to 63]
  Alkaline Phosphatase -Day 70: number analyzed (Participants) | 12 | 13
  Alkaline Phosphatase -Day 70 | 64 [55.5 to 69.5] | 61 [56 to 63]
  Alkaline Phosphatase -Day 182: number analyzed (Participants) | 13 | 14
  Alkaline Phosphatase -Day 182 | 61 [51 to 67] | 64 [51 to 69]
  Alkaline Phosphatase -Day 273: number analyzed (Participants) | 13 | 13
  Alkaline Phosphatase -Day 273 | 63 [57 to 74] | 60 [52 to 68]

5. Primary Outcome: Chemistry and Hematology Laboratory Measures - Creatinine in mg/dL
Description: as for outcome 4
Time Frame: Measured during screening, Days 14, 70, 182, 273
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Group 1: Vaccine | Group 2: Vaccine
Number analyzed (Participants) | 15 | 15
mg/dL
  Creatinine -Baseline | 0.91 [0.8 to 0.98] | 0.79 [0.74 to 0.99]
  Creatinine -Day 14 | 0.89 [0.8 to 0.98] | 0.88 [0.74 to 0.99]
  Creatinine -Day 70: number analyzed (Participants) | 12 | 13
  Creatinine -Day 70 | 0.87 [0.8 to 0.94] | 0.84 [0.81 to 1.04]
  Creatinine -Day 182: number analyzed (Participants) | 13 | 14
  Creatinine -Day 182 | 0.88 [0.86 to 0.97] | 0.82 [0.71 to 0.96]
  Creatinine -Day 273: number analyzed (Participants) | 13 | 13
  Creatinine -Day 273 | 0.91 [0.85 to 0.98] | 0.85 [0.74 to 1]

6. Primary Outcome: Chemistry and Hematology Laboratory Measures - Hemoglobin in g/dL
Description: as for outcome 4
Time Frame: Measured during screening, Days 14, 70, 182, 273
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: g/dL
Arm/Group | Group 1: Vaccine | Group 2: Vaccine
Number analyzed (Participants) | 15 | 15
g/dL
  Hemoglobin -Baseline | 14 [13 to 16] | 14 [13 to 15]
  Hemoglobin -Day 14 | 13 [12 to 15] | 13 [12 to 15]
  Hemoglobin -Day 70: number analyzed (Participants) | 12 | 13
  Hemoglobin -Day 70 | 14 [13 to 16] | 14 [12 to 15]
  Hemoglobin -Day 182: number analyzed (Participants) | 13 | 14
  Hemoglobin -Day 182 | 14 [13 to 16] | 14 [13 to 15]
  Hemoglobin -Day 273: number analyzed (Participants) | 13 | 13
  Hemoglobin -Day 273 | 15 [13 to 15] | 14 [13 to 15]

7. Primary Outcome: Chemistry and Hematology Laboratory Measures - Lymphocyte Count, Neutrophil Count, Platelets, WBC in 1000 Cells/Cubic mm
Description: as for outcome 4
Time Frame: Measured during screening, Days 14, 70, 182, 273
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: 1000 cells/cubic mm
Arm/Group | Group 1: Vaccine | Group 2: Vaccine
Number analyzed (Participants) | 15 | 15
1000 cells/cubic mm
  WBC -Baseline | 6.3 [5.4 to 8.1] | 6.6 [6.3 to 7.8]
  WBC -Day 14 | 6.3 [5.4 to 7.2] | 6.2 [5.2 to 7.6]
  WBC -Day 70: number analyzed (Participants) | 12 | 13
  WBC -Day 70 | 6.4 [5.45 to 7] | 6.3 [4.9 to 7.2]
  WBC -Day 182: number analyzed (Participants) | 13 | 14
  WBC -Day 182 | 6.8 [5.2 to 7.3] | 6.4 [5.3 to 7.9]
  WBC -Day 273: number analyzed (Participants) | 13 | 13
  WBC -Day 273 | 6.2 [5.6 to 7.4] | 6.3 [5.5 to 7]
  Platelets -Baseline | 238 [220 to 316] | 268 [230 to 332]
  Platelets -Day 14 | 257 [220 to 313] | 267 [241 to 352]
  Platelets -Day 70: number analyzed (Participants) | 12 | 13
  Platelets -Day 70 | 238 [214 to 328.5] | 262 [227 to 351]
  Platelets -Day 182: number analyzed (Participants) | 13 | 14
  Platelets -Day 182 | 243 [221 to 311] | 267.5 [232 to 347]
  Platelets -Day 273: number analyzed (Participants) | 13 | 13
  Platelets -Day 273 | 238 [205 to 323] | 265 [236 to 290]
  Lymphocytes -Baseline | 2.128 [1.687 to 2.3] | 2.2 [1.65 to 2.411]
  Lymphocytes -Day 14 | 1.84 [1.39 to 2.118] | 1.98 [1.59 to 2.461]
  Lymphocytes -Day 70: number analyzed (Participants) | 12 | 13
  Lymphocytes -Day 70 | 1.981 [1.619 to 2.317] | 1.91 [1.553 to 2.221]
  Lymphocytes -Day 182: number analyzed (Participants) | 13 | 14
  Lymphocytes -Day 182 | 2.06 [1.7 to 2.55] | 1.874 [1.717 to 2.14]
  Lymphocytes -Day 273: number analyzed (Participants) | 13 | 13
  Lymphocytes -Day 273 | 2.07 [1.879 to 2.198] | 1.729 [1.52 to 1.96]
  Neutrophils -Baseline | 3.74 [2.81 to 5.06] | 3.713 [3.237 to 4.53]
  Neutrophils -Day 14 | 3.631 [2.917 to 4.26] | 3.93 [2.746 to 5.1]
  Neutrophils -Day 70: number analyzed (Participants) | 12 | 13
  Neutrophils -Day 70 | 3.503 [2.923 to 4.32] | 3.437 [2.81 to 4.498]
  Neutrophils -Day 182: number analyzed (Participants) | 13 | 14
  Neutrophils -Day 182 | 3.623 [2.774 to 4.44] | 3.582 [2.825 to 4.684]
  Neutrophils -Day 273: number analyzed (Participants) | 13 | 13
  Neutrophils -Day 273 | 3.329 [2.915 to 5.11] | 3.6 [3.39 to 4.445]

8. Primary Outcome: The Number (Percentage) of Participants With Lab Grade > 1 for ALT, AST, ALP, Creatinine, Hemoglobin, Lymphocyte Count, Neutrophil Count, Platelets, WBC Was Summarized by Arm
Description: The number (percentage) of participants with lab grade > 1 for alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), creatinine, hemoglobin, lymphocyte count, neutrophil count, platelets, white blood cells (WBC) was summarized by arm
Time Frame: Measured during screening, Days 14, 70, 182, 273
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Vaccine | Group 2: Vaccine
Number analyzed (Participants) | 15 | 15
Participants
  Alanine Aminotransferase (U/L)-Baseline | 0 | 0
  Alanine Aminotransferase (U/L)-Day 14 | 0 | 0
  Alanine Aminotransferase (U/L)-Day 70: number analyzed (Participants) | 12 | 13
  Alanine Aminotransferase (U/L)-Day 70 | 0 | 0
  Alanine Aminotransferase (U/L)-Day 182: number analyzed (Participants) | 13 | 14
  Alanine Aminotransferase (U/L)-Day 182 | 0 | 0
  Alanine Aminotransferase (U/L)-Day 273: number analyzed (Participants) | 13 | 13
  Alanine Aminotransferase (U/L)-Day 273 | 0 | 0
  Aspartate Aminotransferase (U/L)-Baseline | 0 | 0
  Aspartate Aminotransferase (U/L)-Day 14 | 0 | 0
  Aspartate Aminotransferase (U/L)-Day 70: number analyzed (Participants) | 12 | 13
  Aspartate Aminotransferase (U/L)-Day 70 | 0 | 0
  Aspartate Aminotransferase (U/L)-Day 182: number analyzed (Participants) | 13 | 14
  Aspartate Aminotransferase (U/L)-Day 182 | 0 | 0
  Aspartate Aminotransferase (U/L)-Day 273: number analyzed (Participants) | 13 | 13
  Aspartate Aminotransferase (U/L)-Day 273 | 0 | 0
  Alkaline Phosphatase (U/L)-Baseline | 0 | 0
  Alkaline Phosphatase (U/L)-Day 14 | 0 | 0
  Alkaline Phosphatase (U/L)-Day 70: number analyzed (Participants) | 12 | 13
  Alkaline Phosphatase (U/L)-Day 70 | 0 | 0
  Alkaline Phosphatase (U/L)-Day 182: number analyzed (Participants) | 13 | 14
  Alkaline Phosphatase (U/L)-Day 182 | 0 | 0
  Alkaline Phosphatase (U/L)-Day 273: number analyzed (Participants) | 13 | 13
  Alkaline Phosphatase (U/L)-Day 273 | 0 | 0
  Hemoglobin (g/dL)-Baseline | 0 | 0
  Hemoglobin (g/dL)-Day 14 | 0 | 0
  Hemoglobin (g/dL)-Day 70: number analyzed (Participants) | 12 | 13
  Hemoglobin (g/dL)-Day 70 | 0 | 0
  Hemoglobin (g/dL)-Day 182: number analyzed (Participants) | 13 | 14
  Hemoglobin (g/dL)-Day 182 | 0 | 0
  Hemoglobin (g/dL)-Day 273: number analyzed (Participants) | 13 | 13
  Hemoglobin (g/dL)-Day 273 | 0 | 0
  Creatinine (mg/dL)-Baseline | 0 | 0
  Creatinine (mg/dL)-Day 14 | 0 | 0
  Creatinine (mg/dL)-Day 70: number analyzed (Participants) | 12 | 13
  Creatinine (mg/dL)-Day 70 | 0 | 0
  Creatinine (mg/dL)-Day 182: number analyzed (Participants) | 13 | 14
  Creatinine (mg/dL)-Day 182 | 0 | 0
  Creatinine (mg/dL)-Day 273: number analyzed (Participants) | 13 | 13
  Creatinine (mg/dL)-Day 273 | 0 | 0
  WBC (1000 cells/cubic mm)-Baseline | 0 | 0
  WBC (1000 cells/cubic mm)-Day 14 | 0 | 0
  WBC (1000 cells/cubic mm)-Day 70: number analyzed (Participants) | 12 | 13
  WBC (1000 cells/cubic mm)-Day 70 | 0 | 0
  WBC (1000 cells/cubic mm)-Day 182: number analyzed (Participants) | 13 | 14
  WBC (1000 cells/cubic mm)-Day 182 | 0 | 0
  WBC (1000 cells/cubic mm)-Day 273: number analyzed (Participants) | 13 | 13
  WBC (1000 cells/cubic mm)-Day 273 | 0 | 0
  Platelets (1000 cells/cubic mm)-Baseline | 0 | 0
  Platelets (1000 cells/cubic mm)-Day 14 | 0 | 0
  Platelets (1000 cells/cubic mm)-Day 70: number analyzed (Participants) | 12 | 13
  Platelets (1000 cells/cubic mm)-Day 70 | 0 | 0
  Platelets (1000 cells/cubic mm)-Day 182: number analyzed (Participants) | 13 | 14
  Platelets (1000 cells/cubic mm)-Day 182 | 0 | 0
  Platelets (1000 cells/cubic mm)-Day 273: number analyzed (Participants) | 13 | 13
  Platelets (1000 cells/cubic mm)-Day 273 | 0 | 0
  Lymphocytes (1000 cells/cubic mm)-Baseline | 0 | 0
  Lymphocytes (1000 cells/cubic mm)-Day 14 | 0 | 0
  Lymphocytes (1000 cells/cubic mm)-Day 70: number analyzed (Participants) | 12 | 13
  Lymphocytes (1000 cells/cubic mm)-Day 70 | 0 | 0
  Lymphocytes (1000 cells/cubic mm)-Day 182: number analyzed (Participants) | 13 | 14
  Lymphocytes (1000 cells/cubic mm)-Day 182 | 0 | 0
  Lymphocytes (1000 cells/cubic mm)-Day 273: number analyzed (Participants) | 13 | 13
  Lymphocytes (1000 cells/cubic mm)-Day 273 | 0 | 0
  Neutrophils (1000 cells/cubic mm)-Baseline | 0 | 0
  Neutrophils (1000 cells/cubic mm)-Day 14 | 0 | 0
  Neutrophils (1000 cells/cubic mm)-Day 70: number analyzed (Participants) | 12 | 13
  Neutrophils (1000 cells/cubic mm)-Day 70 | 0 | 0
  Neutrophils (1000 cells/cubic mm)-Day 182: number analyzed (Participants) | 13 | 14
  Neutrophils (1000 cells/cubic mm)-Day 182 | 0 | 0
  Neutrophils (1000 cells/cubic mm)-Day 273: number analyzed (Participants) | 13 | 13
  Neutrophils (1000 cells/cubic mm)-Day 273 | 0 | 0

9. Primary Outcome: Adverse Events of Special Interest (AESIs)
Description: AEs of special interest (AESI) for this protocol include but are not limited to potential immune-mediated diseases. AESI are reported regardless of relationship to study product(s). All AEs are graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1, July 2017.
Time Frame: Adverse Events of Special Interest (AESI) health contact is at month 18
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Vaccine | Group 2: Vaccine
Number analyzed (Participants) | 15 | 15
Participants
  Y | 0 | 1
  N | 15 | 14

10. Primary Outcome: Occurrence of HIV-specific Total IgG Binding Antibody Response Elicited by the CH505TF gp120 Proteins Produced Via Transient and Stable Transfection Methods Against the Homologous Proteins
Description: Serum HIV-1 specific IgG responses were measured on a BioPlex instrument using a standardized custom HIV1 Luminex assay. The readout was background-subtracted mean fluorescence intensity (MFI). Samples were titrated for IgG to CH505TF gp120 (transient transfection) and CH505TF gp120 (stable transfection) at month 0 (Visit 2) and month 6.5 (Visit 7), with a starting 1:50 dilution followed by a 5-fold dilution series. Net MFI less than 1 is set to 1, and net MFI > 22,000 is set to 22,000. Data are excluded if blood draw date was outside the allowable window, a participant was HIV-infected, reference antigen > 5,000 MFI, or baseline net MFI > 6,500. Samples from post-enrollment visits have positive responses if: (1) the net MFI (MFI minus Blank) values were ≥ antigen-specific cutoff at the 1:50 dilution level for IgG, (2) the net MFI values were greater than 3 times the baseline (day 0) net MFI, and (3) the MFI values were greater than 3 times the baseline MFI values.
Time Frame: Measured at Month 6.5
Population: "Overall number of participants analyzed" represents the HIV uninfected participants with available BAMA data at Month 6.5.
  "Number Analyzed" shows the number of positive responders with available BAMA data after filtering for assay specific quality control criteria at Month 6.5.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Vaccine | Group 2: Vaccine
Number analyzed (Participants) | 13 | 14
Participants
  CH505TF gp120 Stable | 12 | 13
  CH505TF gp120 Transient | 12 | 13

11. Primary Outcome: Levels of HIV-specific Total IgG Binding Antibody Response Elicited by the CH505TF gp120 Proteins Produced Via Transient and Stable Transfection Methods Against the Homologous Proteins (Measured by Net MFI)
Description: Serum HIV-1 specific IgG responses were measured on a BioPlex instrument using a standardized custom HIV1 Luminex assay. The readout was background-subtracted mean fluorescence intensity (MFI), where background referred to a plate level control (i.e., a blank well run on each plate). Net MFI less than 1 is set to 1, and net MFI > 22,000 is set to 22,000. Data are excluded if blood draw date was outside the allowable window, a participant was HIV-infected, reference antigen > 5,000 MFI, or baseline net MFI > 6,500. Samples from post-enrollment visits have positive responses if: (1) the net MFI (MFI minus Blank) values were ≥ antigen-specific cutoff at the 1:50 dilution level for IgG, (2) the net MFI values were greater than 3 times the baseline (day 0) net MFI, and (3) the MFI values were greater than 3 times the baseline MFI values.
Time Frame: Measured at Month 6.5
Population: "Overall number of participants analyzed" represents the number of participants with positive total IgG Binding Antibody responses at Month 6.5.
  "Number Analyzed" shows the number of participants with positive total IgG Binding Antibody responses after filtering for assay specific quality control criteria at Month 6.5.
Measure: Median (Inter-Quartile Range); unit: Net mean fluorescent intensity (net MFI)
Arm/Group | Group 1: Vaccine | Group 2: Vaccine
Number analyzed (Participants) | 12 | 13
Net mean fluorescent intensity (net MFI)
  CH505TF gp120 Stable | 22000 [22000 to 22000] | 22000 [22000 to 22000]
  CH505TF gp120 Transient | 22000 [22000 to 22000] | 22000 [22000 to 22000]

12. Primary Outcome: Area Under Titration Curve of HIV-specific Total IgG Binding Antibody Response Elicited by the CH505TF gp120 Proteins Produced Via Transient and Stable Transfection Methods Against the Homologous Proteins
Description: Samples were titrated for IgG to CH505TF gp120 (transient transfection) and CH505TF gp120 (stable transfection) at month 0 (Visit 2) and month 6.5 (Visit 7), with a starting 1:50 dilution followed by a 5-fold dilution series, ending at 1:156250 dilution. The AUC value was calculated using the trapezoidal rule based on the raw MFI values truncated at zero across the log base 10 dilution series. For each combination of individual and antigen, AUC at each time point was the sum of the areas of the trapezoids calculated between any non-excluded data points in the analyte/titration. AUC was not calculated for any samples which were incompletely titrated, or where a dilution was missing due to failing QC criteria. Data are excluded if blood draw date was outside the allowable window, a participant was HIV-infected, reference antigen > 5,000 MFI, or baseline net MFI > 6,500.
Time Frame: Measured at Month 6.5
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: MFI*log10(1/dilution)
Arm/Group | Group 1: Vaccine | Group 2: Vaccine
Number analyzed (Participants) | 12 | 13
MFI*log10(1/dilution)
  CH505TF gp120 Stable | 21550.9 [16359.2 to 29267.1] | 34973.9 [19147.8 to 39506.9]
  CH505TF gp120 Transient | 23190.6 [18054.6 to 30777.6] | 36942.1 [21130.4 to 43019.9]

13. Secondary Outcome: Occurrence of Neutralizing Antibody (nAB) Response Against CH505TF gp120 Proteins Produced Via Transient and Stable Transfection Methods
Description: Neutralizing antibodies against tier 1 and tier 2 strains of HIV-1 were measured as a function of reductions in Tatregulated luciferase (Luc) reporter gene expression in TZMbl cells. Response to a virus/isolate was considered positive if the neutralization titer was above a prespecified cutoff. A titer was defined as the serum dilution that reduced relative luminescence units (RLUs) by 50% and 80% relative to the RLUs in virus control wells (cells + virus only) after subtraction of background RLU (cells only). The prespecified cutoff for ID50 and ID80 was 10. Data are excluded if blood draw date was outside the allowable window, assay results are deemed unreliable for analysis by the lab, or a participant was HIV-infected.
Time Frame: Measured at Months 2.5 and 6.5
Population: "Overall number of participants analyzed" represents the HIV uninfected participants with available nAB data at Months 2.5 and/or 6.5.
  "Number Analyzed" shows the number of HIV uninfected participants with available nAB data after filtering for assay specific quality control criteria at each timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Vaccine | Group 2: Vaccine
Number analyzed (Participants) | 14 | 14
Participants
  CH505.w4.3, Titer, (ID50), V5, M2.5: number analyzed (Participants) | 12 | 13
  CH505.w4.3, Titer, (ID50), V5, M2.5 | 11 | 13
  CH505.w4.3, Titer (ID50), V7, M6.5: number analyzed (Participants) | 13 | 14
  CH505.w4.3, Titer (ID50), V7, M6.5 | 12 | 14
  CH505.w4.3, Titer (ID80), V5, M2.5: number analyzed (Participants) | 12 | 13
  CH505.w4.3, Titer (ID80), V5, M2.5 | 10 | 12
  CH505.w4.3, Titer (ID80), V7, M6.5: number analyzed (Participants) | 13 | 14
  CH505.w4.3, Titer (ID80), V7, M6.5 | 11 | 13
  CH505TF, Titer (ID50), V5, M2.5: number analyzed (Participants) | 12 | 13
  CH505TF, Titer (ID50), V5, M2.5 | 0 | 0
  CH505TF, Titer (ID50), V7, M6.5: number analyzed (Participants) | 13 | 14
  CH505TF, Titer (ID50), V7, M6.5 | 0 | 2
  CH505TF, Titer (ID80), V5, M2.5: number analyzed (Participants) | 12 | 13
  CH505TF, Titer (ID80), V5, M2.5 | 0 | 0
  CH505TF, Titer (ID80), V7, M6.5: number analyzed (Participants) | 13 | 14
  CH505TF, Titer (ID80), V7, M6.5 | 0 | 0

14. Secondary Outcome: Neutralization Titers of nAB Responses Against CH505TF gp120 Proteins Produced Via Transient and Stable Transfection Methods
Description: Neutralizing antibodies against tier 1 and tier 2 strains of HIV-1 were measured as a function of reductions in Tatregulated luciferase (Luc) reporter gene expression in TZMbl cells. Response magnitudes were assessed using neutralization titer, which is defined as the serum dilution that reduced relative luminescence units (RLUs) by 50% and 80% relative to the RLUs in virus control wells (cells + virus only) after subtraction of background RLU (cells only). Higher neutralization titer indicates higher response level. Response to a virus/isolate was considered positive if the neutralization titer was above 10. Data are excluded if blood draw date was outside the allowable window, assay results are deemed unreliable for analysis by the lab, or a participant was HIV-infected.
Time Frame: Measured at Months 2.5 and 6.5
Population: "Overall number of participants analyzed" represents the number of participants with positive nAB responses at Months 2.5 and/or 6.5.
  "Number Analyzed" shows the number of participants with positive nAB responses after filtering for assay specific quality control criteria at each timepoint.
Measure: Median (Inter-Quartile Range); unit: 1/dilution
Arm/Group | Group 1: Vaccine | Group 2: Vaccine
Number analyzed (Participants) | 13 | 14
1/dilution
  CH505.w4.3, Titer (ID50), V5, M2.5: number analyzed (Participants) | 11 | 13
  CH505.w4.3, Titer (ID50), V5, M2.5 | 135.7 [72.8 to 226.7] | 122.9 [68.8 to 185.1]
  CH505.w4.3, Titer (ID50), V5, M6.5: number analyzed (Participants) | 12 | 14
  CH505.w4.3, Titer (ID50), V5, M6.5 | 492.5 [144.7 to 1126.3] | 404.1 [219.9 to 1274.9]
  CH505.w4.3, Titer (ID80), V7, M2.5: number analyzed (Participants) | 10 | 12
  CH505.w4.3, Titer (ID80), V7, M2.5 | 32.9 [24.6 to 56.5] | 39.4 [25.5 to 55.8]
  CH505.w4.3, Titer (ID80), V7, M6.5: number analyzed (Participants) | 11 | 13
  CH505.w4.3, Titer (ID80), V7, M6.5 | 173.2 [77.4 to 300.8] | 135.7 [77 to 356.7]
  CH505TF, Titer (ID50), V5, M2.5: number analyzed (Participants) | 0 | 0
  CH505TF, Titer (ID50), V5, M6.5: number analyzed (Participants) | 0 | 2
  CH505TF, Titer (ID50), V5, M6.5 |  | 11.6 [11.5 to 11.7]
  CH505TF, Titer (ID80), V7, M2.5: number analyzed (Participants) | 0 | 0
  CH505TF, Titer (ID80), V7, M6.5: number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Serious Adverse events and non-serious adverse are collected until month 12. All-cause mortality are collected until month 18.
Arm/Group | Group 1: Vaccine | Group 2: Vaccine
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 1/15 | 0/15
Other Adverse Events (participants affected / at risk) | 7/15 | 7/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Vaccine (N=15) | Group 2: Vaccine (N=15)
Any Event in SOC (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Vaccine (N=15) | Group 2: Vaccine (N=15)
Any Event in SOC (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Any Event in SOC (General disorders) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Any Event in SOC (Infections and infestations) | 3 (3) | 5 (5)
Influenza (Infections and infestations) | 1 (1) | 2 (2)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Any Event in SOC (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Any Event in SOC (Investigations) | 3 (6) | 3 (3)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood creatine increased (Investigations) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 3 (3) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1)
Any Event in SOC (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Any Event in SOC (Nervous system disorders) | 1 (1) | 0 (0)
Sensory disturbance (Nervous system disorders) | 1 (1) | 0 (0)
Any Event in SOC (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Any Event in SOC (Vascular disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol (2018-12-12): https://cdn.clinicaltrials.gov/large-docs/96/NCT03856996/Prot_003.pdf
  • Statistical Analysis Plan: Safety SAP (2019-07-23): https://cdn.clinicaltrials.gov/large-docs/96/NCT03856996/SAP_002.pdf
  • Statistical Analysis Plan: Immunogenicity SAP (2023-08-21): https://cdn.clinicaltrials.gov/large-docs/96/NCT03856996/SAP_004.pdf
  • Informed Consent Form (2019-05-14): https://cdn.clinicaltrials.gov/large-docs/96/NCT03856996/ICF_000.pdf